CLINICAL TRIAL: NCT01651273
Title: A Site and Subject Blinded Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS 852927 in Patients With Primary Hypercholesterolemia on a Stable Dose of Statin Therapy
Brief Title: A Safety Study of BMS-852927 in Subjects With Hypercholesterolemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV201-008; 2012-001946-17 (EudraCT Number)
Record Dates: First submitted 2012-07-13; First posted 2012-07-27 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: BMS-852927 (0.25 mg) (Experimental)
  Interventions: Drug: BMS-852927
- Arm 2: BMS-852927 (1.0 mg) (Experimental)
  Interventions: Drug: BMS-852927
- Arm 3: BMS-852927 (2.5 mg) (Experimental)
  Interventions: Drug: BMS-852927
- Arm 4: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-852927 — Capsules, Oral, 0.25 mg, Once daily, 28 days
  Arms: Arm 1: BMS-852927 (0.25 mg)
Drug: BMS-852927 — Capsules, Oral, 1.0 mg, Once daily, 28 days
  Arms: Arm 2: BMS-852927 (1.0 mg)
Drug: BMS-852927 — Capsules, Oral, 2.5 mg, Once daily, 28 days
  Arms: Arm 3: BMS-852927 (2.5 mg)
Drug: Placebo — Capsules, Oral, 0 mg, Once daily, 28 days
  Arms: Arm 4: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of BMS-852927 after 28 days of dosing in patients with high cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged ≥18 to ≤75
* Body mass index (BMI) ≤ 40 kg/m2
* Primary hypercholesterolemia on a stable daily dose of a statin for ≥ 6 weeks
* Serum triglyceride levels at screening < 400mg/dL (< 4.52 mmol/L)

Exclusion Criteria:

* Any significant acute medical illness, significant cardiovascular history
* Current or history of hepatic or hepatobiliary disease
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number and percent of subjects that experience the Serious adverse events, Deaths, Adverse events leading to discontinuation of study therapy | Up to 56 days of study participation
Number and percent of subjects that experience the Serious adverse events, Deaths, Adverse events leading to discontinuation of study therapy | Up to 30 days post discontinuation of dosing or last participation in the study for serious adverse events collection
Number and percent of subjects with potentially clinically significant changes in ECG parameter | Upto 56 days
  Electrocardiogram (ECG) parameters defined as:
  * Investigator identified clinically significant abnormalities
  * QTcF> 480 msec or QTcF changes from baseline> 60 msec
  * QRS (msec): QRS> 120 msec
  * PR (msec): PR > 210 msec
Number and percent of subjects with potentially clinically significant changes in low density lipoprotein (LDL)-c (measured) | Upto 56 days
  LDL-c (measured) defined as:
  * LDL-c (mg/dL): LDL-c percent changes from baseline >= 15%

SECONDARY OUTCOMES:
Trough observed concentration (Cmin) of BMS-852927 will be derived from plasma concentration versus time data | Days 7, 14, 21 and 28
Area under the concentration-time curve from zero (pre-dose) to 8 h [AUC(0-8h)] of BMS-852927 will be derived from plasma concentration versus time data | Days 1 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- Canada (5):
  - Local Institution, Brampton, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Pointe-Claire, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution, Victoriaville, Quebec
- Germany (2):
  - Local Institution, Berlin
  - Local Institution, Neuss

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx